CLINICAL TRIAL: NCT01590914
Title: Brain Activation in Response to Appetite Cues Pre- and Post- Bariatric Surgery
Brief Title: Brain Activation in Response to Appetitive Cues Pre- and Post- Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Obesity and Nutrition Research Center (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Dr. Allan Geliebter, Principal Investigator, New York Obesity and Nutrition Research Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 08-174
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: Roux-en-Y Bariatric surgery,; Gastric banding,; fMRI,; food cues
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Roux-En Y Gastric Bypass (Experimental): 40 subjects who plan to undergo Roux-En-Y Gastric Bypass bariatric surgery. BOLD fMRI responses to food cues will be collected in the Fed Condition and Fasted Condition Pre-Surgery and 3 months post Surgery.
  Interventions: Procedure: Fed Condition; Procedure: Fasted Condition
- Gastric Banding (Experimental): 40 Subjects who plan to undergo Gastric Banding bariatric Surgery. BOLD fMRI responses to food cues will be collected in the Fed Condition and Fasted Condition Pre-Surgery and 3 months post Surgery.
  Interventions: Procedure: Fed Condition; Procedure: Fasted Condition
- Formula Diet Weight-Loss (Experimental): 40 subjects will undertake a 12-week liquid formula weight loss plan. BOLD fMRI responses to food cues will be collected in the Fed Condition and Fasted Condition pre-weight loss and 3 months after a 12-week weight loss plan.
  Interventions: Procedure: Fed Condition; Procedure: Fasted Condition
- No Treatment (Experimental): 40 subjects who do not undergo any treatment for weight loss. BOLD fMRI responses to food cues will be collected in the Fed Condition and Fasted Condition at baseline and after 3 months.
  Interventions: Procedure: Fed Condition; Procedure: Fasted Condition

INTERVENTIONS:
Procedure: Fed Condition — Subjects will consume a 250ml liquid test meal (250kcal) before undergoing a 40min fMRI scan to assess the BOLD signal responses to visual and auditory responses to food and non-food cues.
Procedure: Fasted Condition — Subjects will consume a 250ml control (water) before undergoing a 40min fMRI scan to assess BOLD signal response to visual and auditory food and non-food cues

SUMMARY:
Utilizing fMRI, this study will examine changes in BOLD signal as a proxy measure of brain activation in response to highly palatable (high energy density [kcal/g]), less palatable and non-food stimuli in severely obese women pre, 1 month post and 3 months post undergoing bariatric surgery (in surgery patients) and at equivalent times for control groups in fed and fasted conditions at each time point.

Two surgical groups: (i) laparoscopic Roux-en-Y gastric bypass (RYGB) and (ii) gastric banding (GB) will be compared with two control groups: (i)those enrolled on a 3-month formula weight loss program or (ii) those who qualify, but do not undergo bariatric surgery, and receive no weight loss treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 65 years
* BMI > 40 and < 50kg/m2
* Right handed
* Good comprehension of English

Exclusion Criteria:

* > 5% weight fluctuation in the past 3 months
* Presence of disease (including diabetes)
* Pregnancy, lactation or planning to become pregnant in next 18mon
* Smoking, or or recent (within past 12 month) smoking cessation
* Consumption of > 3 alcoholic beverages per day
* Left handed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
BOLD signal response to visual and auditory food cues | pre-surgery, 1mo post and 3mo post surgery
  BOLD signal changes in the brain in response to highly palatable (high energy density [kcal/g]), less palatable (low energy density)and non-food, stimuli in severely obese women pre-surgery, 1 month post-surgery and 3 months post bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Allan Geliebter, PhD, Principal Investigator — New York Nutrition & Obesity Research Center
Locations (2):
- United States (2):
  - St Luke's Roosevelt Hospital Center, New York, New York
  - Columbia University Medical Center, New York, New York